CLINICAL TRIAL: NCT03305666
Title: A Randomized Clinical Trial of Single Dose Liposomal Bupivacaine Delivered Via VATS Intercostal Nerve Block vs. Continuous Bupivacaine Infusion Delivered Via Indwelling Subscapular Catheter After Surgical Stabilization of Rib Fractures
Brief Title: Trial of Injected Liposomal Bupivacaine vs Bupivacaine Infusion After Surgical Stabilization of Rib Fractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-0685
Record Dates: First submitted 2017-10-04; First posted 2017-10-10 (Actual); Results first posted 2021-08-25 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Drug Effect; Rib Fractures; Rib Trauma; Surgical Procedure, Unspecified; Pain; Catheter (Other); Nerve Pain; Local Infiltration; Anesthesia, Local; Intercostal Rib; Opioid Dependence; Chest Injury Trauma; Pneumonia
MeSH Terms: conditions — Rib Fractures; Pain; Neuralgia; Opioid-Related Disorders; Pneumonia

STUDY DESIGN:
Intervention Model Description: Non-inferiority, randomized, clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bupivacaine indwelling catheter (Active Comparator): Bupivacaine indwelling OnQ pain pump catheter will be placed in the subscapular space at the time of surgery, at infusion of 12 ml/hr of 0.25% bupivacaine, and left in place for a maximum of 120 hours
  Interventions: Drug: Bupivacaine indwelling catheter
- Liposomal bupivacaine injection (Active Comparator): A single injection of liposomal bupivacaine: mixture of 20 mL liposomal bupivacaine, 20 mL 0.25% bupivacaine, and 10 mL sterile saline (50 mL total), will be delivered in the intercostal space during VATS (with a 178 mm, 22 gauge needle, at ribs 3-8).
  Interventions: Drug: Liposomal bupivacaine injection

INTERVENTIONS:
Drug: Liposomal bupivacaine injection — A single injection of liposomal bupivacaine is administered at the time of SSRF, directly to the fracture site via VATS
  Other Names: Exparel
  Arms: Liposomal bupivacaine injection
Drug: Bupivacaine indwelling catheter — Bupivacaine indwelling OnQ pain pump catheter is placed in the subscapular space at the time of SSRF for continuous bupivacaine infusion post op
  Other Names: OnQ pain pump, Continuous infusion of bupivacaine
  Arms: Bupivacaine indwelling catheter

SUMMARY:
Rib fractures represent a common injury pattern this is highly associated with patient morbidity and mortality, as pain control remains a challenge. Even after surgical stabilization of rib fractures (SSRF), unsuccessful pain control can lead to morbid outcomes such as pneumonia and opioid dependence. Multi-modal anesthesia, with the use of thoracic epidurals and para-vertebral injections/catheters, has shown to lessen these occurrences but are subject to a wide array of limitations. A more directed therapy with liposomal bupivacaine has shown to provide sustained analgesia for up to 72 hours in patients who have undergone other types of thoracic surgery, but not SSRF. The hypothesis of the current clinical trial is that, among patients undergoing SSRF, liposomal bupivacaine delivered via video assisted thoracic surgery (VATS) is an intercostal nerve block that provides comparable analgesia to the pain catheter, as measured by pulmonary function, numeric pain scoring, and postoperative narcotic use.

DETAILED DESCRIPTION:
Rib fractures represent a common injury pattern with high associated morbidity and mortality. Effective pain control in both the acute and long term periods remains a challenge. Surgical stabilization of rib fractures (SSRF) is now a recommended treatment for patients with severe chest wall injuries. In addition to stabilization of the chest wall, SSRF offers a unique opportunity to deliver directed, loco-regional anesthesia. Loco-regional anesthesia is a recognized, essential component of multi-modal anesthesia for patients with rib fractures in order to both decrease pain and minimize the use of opioids and their associated side effects.

Delivery options for loco-regional anesthesia to patients with rib fractures share in common the intention of anesthetizing the intercostal nerves. Moving from the spinal cord laterally, modalities include thoracic epidural catheters, paravertebral blocks or catheters, and rib/intercostal blocks. Although rib blocks may be accomplished via a variety of techniques, the two most common intra-operative techniques are video-assisted thoracoscopic surgery (VATS) intercostal nerve blocks and indwelling, subscapular catheters In general, neuraxial modalities such as thoracic epidural and para-vertebral injections/catheters are subject to a wide array of limitations, including patient coagulopathy (International Normalized Ratio > 1.5), co-existing spine fractures, peri-insertion, peri-removal withholding of venous thromboembolism pharmacoprophylaxis, and provider availability. For these reasons, our current practice is to insert a subscapular "pain catheter" at the conclusion of the SSRF operation; this catheter is able to deliver a continuous infusion of 0.25% bupivacaine and may be left in place for several days.

Although favorable results using the pain catheter have been published in patients with rib fractures who have not undergone SSRF, we have noticed several limitations to this treatment modality. First, position is highly variable; and, because the catheter is not truly in the space of the intercostal nerves, drug delivery is likely irregular. This variability may be particularly relevant in obese patients; and the median body mass index of patient who underwent SSRF at Denver Health is 29 kg/m^2. Beyond catheter placement, we have also experienced issues with leakage of drug from the skin entry site of the catheter. Moreover, catheters frequently become dislodged or inadvertently removed during patient transport. Further, the indwelling foreign body likely introduces some risk of infection. Finally, the presence of the catheter is distressing to many patients.

Liposomal bupivacaine (Exparel, Pacira Pharmaceuticals, Inc., Parsippany, NJ, www.pacira.com) has been shown to provide sustained analgesia for up to 72 hours following a single injection of the drug delivery system. The safety and efficacy of liposomal bupivacaine has been evaluated in over 1,300 subjects and 21 clinical trials. Although many of these trials have included thoracic surgery patients, no trial has evaluated the efficacy and safety of liposomal bupivacaine administered to patients with rib fractures undergoing SSRF. Potential benefits as compared to current practice include directed injection immediately adjacent to the intercostal nerve using a VATS approach, as well as obviation of the need for an indwelling catheter. The hypothesis of the current clinical trial is that, among patients undergoing SSRF, liposomal bupivacaine delivered via video assisted thoracic surgery (VATS) is an intercostal nerve block that provides comparable analgesia to the pain catheter, as measured by pulmonary function, numeric pain scoring, and postoperative narcotic use.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing SSRF at Denver Health Medical Center

Exclusion Criteria:

* Allergy or hypersensitivity to bupivacaine
* Pregnancy
* Incarceration
* Age < 18 years
* Indwelling continuous thoracic epidural analgesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fredric Pieracci, MD MPH, Principal Investigator — Denver Health and Hospital
Locations (1):
- Denver Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leasia KN, Ciarallo C, Prins JTH, Preslaski C, Perkins-Pride E, Hardin K, Cralley A, Burlew CC, Coleman JJ, Cohen MJ, Lawless R, Platnick KB, Moore EE, Pieracci FM. A randomized clinical trial of single dose liposomal bupivacaine versus indwelling analgesic catheter in patients undergoing surgical stabilization of rib fractures. J Trauma Acute Care Surg. 2021 Nov 1;91(5):872-878. doi: 10.1097/TA.0000000000003264. PMID 33951024

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral for surgical stabilization of rib fracture (SSRF) at Denver Health from November 2017 through July 2020.
Pre-assignment Details: All 36 patients were enrolled in the study and assigned to groups via a Microsoft Excel randomization.
Period: Overall Study
Arm/Group | Bupivacaine Indwelling Catheter | Liposomal Bupivacaine Injection
Started | 18 | 18
Completed | 16 | 18
Not Completed | 2 | 0
Not completed — ORIF cancelled due to patient's cognitive decline, withdrawn from study at this time | 2 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis did not include two patients who were withdrawn from the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine Indwelling Catheter | Liposomal Bupivacaine Injection | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 15 | 26
  >=65 years | 5 | 3 | 8
Age, Continuous [Mean (Full Range); unit: years] | 53.3 [18 to 81] | 52.3 [37 to 85] | 52.8 [18 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 11 | 10 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 10 | 13 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 16 | 16 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 26 [20.4 to 34.8] | 27.2 [16.45 to 36.8] | 26.6 [16.45 to 36.8]
Injury Severity Score (ISS) [Mean (Full Range); unit: units on a scale] — The total range of the Injury Severity Score (ISS) is from 0-75, with a score of 0 being the best and indicating no injury at all and a score of 75 being the worst and indicating a fatal injury. Six major body regions are scored by a physician on a scale of 0-6 and the body regions with the three most severe injury scores are squared and summed to result in the final 0-75 score. However, if any of the three scores is a 6, the final score is automatically set at 75.
  units on a scale | 19.5 [9 to 38] | 22.1 [9 to 38] | 20.8 [9 to 38]
Number of Participants with Asthma [Count of Participants; unit: Participants] | 2 | 3 | 5
Number of Participants with COPD [Count of Participants; unit: Participants] | 0 | 0 | 0
Number of Participants who Use Tobacco [Count of Participants; unit: Participants] | 5 | 3 | 8
Admit Glasgow Coma Scale (GCS) [Mean (Full Range); unit: units on a scale] — The Glasgow Coma Scale (GCS) is a measure of consciousness scale examining patients' degree of responsiveness regarding eye opening, verbal communication, and motor functioning. The GCS scores have a range of 3-15, with a 3 being the worst score and a 15 being the best. Eye opening is scored from 1-4, verbal communication is scored from 1-5, and motor functioning is scored from 1-6. The three scored categories are summed to arrive at the total score, averaged across patients below.
  units on a scale | 13.3 [3 to 15] | 13.3 [3 to 15] | 13.3 [3 to 15]

OUTCOME MEASURES:

1. Primary Outcome: Daily Sequential Clinical Assessment of Respiratory Function (SCARF) Score
Description: The SCARF score is a validated, dynamic tool that ranges from 0-4, with 0 being the best score and 4 being the worst. One point is given for each of the following four parameters: (1) respiratory rate ≥ 20 breaths per minute; (2) numeric pain score ≥ 5; (3) incentive spirometry < 50% of predicted based upon a nomogram including sex, height, and age; (4) cough deemed inadequate to clear respiratory secretions by respiratory therapists. The parameters used to calculate the SCARF score are summed to create the total 0-4 score and these results were recorded by clinical personnel not involved in the trial. SCARF scores were taken at 10 am daily for all postoperative inpatient hospital days, however due to variance in length of stay, only scores from the first 5 postoperative days were recorded for the purpose of this results analysis. Scores were then aggregated across the patients and timeframe to result in one median score per group.
Time Frame: Median SCARF scores were recorded for the first 5 postoperative days.
Population: All 34 participants were analyzed on this data point and aggregate data is provided below for each treatment arm. Patients who were intubated at 10 am (the time of data reporting) could not be measured on a few factors of this outcome measure and this discrepancy was accounted for in the statistical analysis.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Bupivacaine Indwelling Catheter | Liposomal Bupivacaine Injection
Number analyzed (Participants) | 16 | 18
score on a scale | 2 [0 to 4] | 2 [0 to 4]
Statistical Analysis 1: Comparison: Bupivacaine Indwelling Catheter vs Liposomal Bupivacaine Injection; Test type: Non-Inferiority — Statistical analyses were conduced using SAS version 9.4. This non-inferiority test was conducted via a one-way ANOVA test, with statistical significance set at p < 0.05; p = 0.12, ANOVA

2. Secondary Outcome: Daily Narcotic Requirements Using Equi-analgesic Doses
Description: Narcotic pain medication requirements were recorded daily over the duration of inpatient hospital stay, however due to variance in length of stay, only the first 5 postoperative days were recorded for this analysis. Scores were averaged across patients providing one daily postoperative mean score per treatment group. The narcotics provided to patients varied based on standard of care, so an Equi-Analgesic Scale was used to standardize dosages across narcotic type. A 1:1 ratio for narcotic dosages is calculated with the following measured as equivalent: 1.5 milligrams (mg) of intravenous (IV) Hydromorphone; 7.5 mg of per oral (PO) Hydromorphone; 100 micrograms (mcg) of IV Fentanyl; 10 mg of IV Morphine; 30 mg of PO Morphine; 20 mg of PO Oxycodone (Percocet); and 30 mg of PO Hydrocodone (Vicodin). In the context of this scale, lower scores are best, indicating fewer narcotics required and higher scores are worse indicating the need for more narcotics based on subjective patient pain.
Time Frame: Mean narcotic requirement scores were recorded for the first 5 postoperative hospital inpatient days.
Population: All 34 participants were analyzed on this data point and aggregate data is provided below for each treatment arm. The data below is the mean result provided for each of the first 5 postoperative days following surgical intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine Indwelling Catheter | Liposomal Bupivacaine Injection
Number analyzed (Participants) | 16 | 18
units on a scale
  Postoperative Day #1 | 8.8 (13) | 6.5 (8.5)
  Postoperative Day #2 | 6.8 (10.1) | 4.0 (6.9)
  Postoperative Day #3 | 4.0 (6.1) | 2.6 (3.3)
  Postoperative Day #4 | 4.2 (5.7) | 1.6 (1.5)
  Postoperative Day #5 | 4.1 (7.4) | 2.2 (2.3)
Statistical Analysis 1: Comparison: Bupivacaine Indwelling Catheter vs Liposomal Bupivacaine Injection; This is the P-Value for between groups comparison of Postoperative Day #1; Test type: Non-Inferiority — Statistical analyses were conducted using SAS version 9.4. This non-inferiority test was conducted via a one-way ANOVA test, with statistical significance set at p < 0.05; p = 0.41, ANOVA
Statistical Analysis 2: Comparison: Bupivacaine Indwelling Catheter vs Liposomal Bupivacaine Injection; This is the P-Value for between groups comparison of Postoperative Day #2; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.25, ANOVA
Statistical Analysis 3: Comparison: Bupivacaine Indwelling Catheter vs Liposomal Bupivacaine Injection; This is the P-Value for between groups comparison of Postoperative Day #3; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.12, ANOVA
Statistical Analysis 4: Comparison: Bupivacaine Indwelling Catheter vs Liposomal Bupivacaine Injection; This is the P-Value for between groups comparison of Postoperative Day #4; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.04, ANOVA
Statistical Analysis 5: Comparison: Bupivacaine Indwelling Catheter vs Liposomal Bupivacaine Injection; This is the P-Value for between groups comparison of Postoperative Day #5; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.32, ANOVA

3. Secondary Outcome: Percentage of Participants Experiencing Failure of Primary Loco-Regional Analgesia (LRA)
Description: The failure of LRA for this study was defined as the percentage number of instances a patient required a secondary LRA modality within 72 hours of placement of the primary modality for either treatment arm. Requirement of this secondary LRA was determined by the patients' medical team with criteria based on subjective patient experience of pain.
Time Frame: 72 hours
Population: All 34 participants were analyzed on this data point and aggregate data is provided below for each treatment arm. Percentages entered below are based on number of failure occurrences, in this case defined as requiring a secondary LRA.
Measure: Number; unit: percentage of participants
Arm/Group | Bupivacaine Indwelling Catheter | Liposomal Bupivacaine Injection
Number analyzed (Participants) | 16 | 18
percentage of participants | 18.8 | 5.6
Statistical Analysis 1: Comparison: Bupivacaine Indwelling Catheter vs Liposomal Bupivacaine Injection; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.23, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the participants' stay in the hospital or for 28 days, whichever length of time was the shorter duration.
Arm/Group | Bupivacaine Indwelling Catheter | Liposomal Bupivacaine Injection
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 3/16 | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine Indwelling Catheter (N=16) | Liposomal Bupivacaine Injection (N=18)
Hospital Readmission (Social circumstances) | 1 (2) | 0 (0) — EtOH Withdrawal; not study related.
Hospital Readmission (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Chronic subdural hematoma requiring evacuation; not study related.
OR Takeback (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Evacuation of incisional hematoma
ED Visit (Social circumstances) | 1 (1) | 0 (0) — Acute EtOH intoxication, complaint of rib pain, however no admission.

LIMITATIONS AND CAVEATS:
There were no limitations that created barriers to the completion of this project. While this was expected at the outset of this exploratory trial, there was a relatively small sample size with a wide range of fractures for individual participants. Underpowering likely limited analyses of secondary outcomes such as narcotic requirements and failure of LRA. The study also excluded patients with GCS < 8, so caution should be exercised when extrapolating to mechanically ventilated patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT03305666/Prot_SAP_000.pdf